CLINICAL TRIAL: NCT01444820
Title: Phase III Study of Hypofractionated, Dose Escalation Radiotherapy for High Risk Adenocarcinoma of the Prostate, Using 3D-CRT or Intensity-Modulated Radiotherapy
Brief Title: Hypofractionated, Dose Escalation Radiotherapy for High Risk Adenocarcinoma of the Prostate
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Tamim Niazi, Radiation Oncologist, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS V
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: radiation therapy; hypofractionation; hormonal therapy; high risk adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation Dose Hypofractionation; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypofractionation (Experimental): One phase technique (IMRT or 3D-CRT): radiotherapy to the prostate + pelvic lymphnodes
  Interventions: Radiation: hypofractionation
- Conventional (Other): two-phase technique (IMRT or 3D-CRT): 1) whole pelvis including the prostate and regional lymph nodes; 2) boost to the prostate
  Interventions: Radiation: conventional

INTERVENTIONS:
Radiation: hypofractionation — Centres using IMRT will use the dose painting technique to treat the prostate + proximal 1-cm SV to 6800 cGy in 25 fractions while the pelvic lymph nodes will receive 4500 cGy in 25 fractions. For patients with T3b, the whole SV is to be treated to 6800 cGy. Institutions using 3D-CRT will deliver the required dose to the pelvic volume (including pelvic lymph nodes and boost volume) - 4500 cGy - and a concomitant boost to the prostate and proximal 1-cm (or the whole SV if involved) SV to 6800 cGy.
  Arms: Hypofractionation
Radiation: conventional — The first phase: whole pelvis including the prostate and regional lymph nodes treated with 4400 cGy in 22 fractions.
  The second phase: prostate + proximal 1-cm SV treated with 3200 cGy in 16 fractions.
  For patients with T3b, the whole SV is to be treated to 7600 cGy.
  Arms: Conventional

SUMMARY:
In North America, around a quarter a million men are diagnosed with prostate cancer every year, and about 31,000 patients will die of their disease each year. Like other western countries, the incidence in Canada has increased due to an aging population and prostate specific antigen (PSA) screening. This has led to a significant demand on cancer care services for these patients. Prostate cancer patient with high risk features are more often treated with external beam radiation therapy (EBRT) plus two to three years of hormonal manipulation (luteinizing hormone-releasing hormone [LHRH] agonist). The most common radiation dose treatment for these patients is 74-78 Gy in 37-39 daily fractions of 180-200 cGy for a treatment length of 7.5 weeks. This fraction size is believed to offer the best balance between desired tumour kill and unwanted normal tissue injury. Larger fraction sizes of more than 250 cGy (hypofractionation) are usually avoided for curative therapy because late reacting normal tissues. However prostate cancer cells have a unique radiobiology characteristic that suggests that hypofractionated radiotherapy is more efficient at prostate tumour killing than standard fractionation is, and will produce equivalent tumour control with a lower total dose and a shorter overall treatment time. Improved target localization techniques and conformal radiation therapy technology have allowed for dose escalation and hypofractionated radiation delivery in these circumstances with minimal or no increased toxicities.

This trial is designed to determine whether high risk prostate cancer patients can be safely treated with a dose escalation hypofractionated radiation therapy in 5 weeks as opposed to the usual 7-8 weeks. These patients will be randomized to either the usual 76 Gy in 38 fractions or 68 Gy in 25 fractions. 3D-Conformal Radiotherapy (3D-CRT) or Intensity Modulated Radiotherapy (IMRT) will be used to deliver the required radiation dose. Patients will also receive 28 months of androgen deprivation therapy (LHRH agonist). The primary outcome of the study is the acute and delayed toxicity and the secondary outcomes include biochemical failure, prostate specific mortality rate, bone metastases free survival, the prognostic and predictive value of several biological variables: presence of the PTEN deletion; expression of FoxP3 gene variants, topoisomerase 2α and cancer testis antigens; expression of X chromosome-linked micro-RNAs; presence of TMRSS2-ERG gene fusion and quality of life. It is planned to recruit 250 patients to this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate diagnosed within 6 months prior to randomization
2. Patient has been classified as high risk defined clinically as: T3 or T4, Gleason Score > 8, and/ or PSA > 20 (ng/mL or μg/L).
3. Pelvic and para-aortic lymph nodes must be negative on computerized tomography (CT scan) or magnetic resonance imaging (MRI) of the abdomen and pelvis performed within 12 weeks prior to randomization.
4. Investigations, including chest X-ray or chest CT scan and bone scan (with radiographs of suspicious areas) have been performed within 12 weeks prior to randomization and are negative for metastases.
5. Patients will have had a PSA test done at the time of diagnosis. This PSA test could be repeated within 28 days prior to randomization.
6. The patient may have received prior androgen suppression therapy provided that androgen suppression therapy commenced no more than 28 days prior to randomization.
7. The patient must not have received any cytotoxic anticancer therapy for prostate cancer prior to randomization.
8. ECOG performance status must be 0 or 1
9. Hematology and biochemistry: should be done within 28 days prior to randomization:

   1. Hemoglobin > 100 g/L
   2. Absolute Neutrophils > 1.5 x 109/L
   3. Platelets > 100 x 109/L
   4. AST and/or ALT < 1.5 x Upper Limit of Normal (ULN)
   5. Alkaline phosphatase < 2.5 x Upper Limit of Normal (ULN)
   6. Total bilirubin < ULN
   7. Serum creatinine < 1.5 x ULN
10. adequate birth control measures should be used by the participant
11. Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements.
12. Patients must be accessible for treatment and follow-up.

Exclusion Criteria:

1. Patients with a history of other malignancies, except: non-melanoma skin cancer; or other solid tumours curatively treated with no evidence of disease for > 5 years.
2. The presence of small-cell or transitional-cell carcinoma in the biopsy specimen.
3. Patients who had previous chemotherapy for carcinoma of the prostate.
4. Patients who had prior surgical treatment for carcinoma of the prostate apart from trans-urethral resection, including bilateral orchiectomy.
5. Patients with any contraindication to pelvic radiotherapy: including, but not limited to, previous pelvic radiotherapy, inflammatory bowel disease or severe bladder irritability.
6. Patients with serious non malignant disease resulting in a life expectancy less than 3 years.
7. Other serious illness, psychiatric or medical condition that would not permit the patient to be managed according to the protocol
8. Known hypersensitivity to any protocol-indicated study medications.
9. Presence of bilateral hip replacement prostheses.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Acute and delayed genito-urinary and gastrointestinal toxicity differences | 6-8 years
  primary outcome is the acute and delayed genito-urinary and gastrointestinal toxicity differences (at or before 90 days for the acute and 90-180 days and after for the delayed toxicity) in high risk prostate cancer patients treated with the hypofractionation vs standard of care regimen using 3D-CRT or IMRT.

SECONDARY OUTCOMES:
freedom from biochemical failure | 3 years and 5 years post-treatment
  To measure freedom from biochemical failure at 3 and 5 years.
disease free and overall survival | at 5 years
  To measure disease specific and overall survival at 5 years
Correlation of rectum and bladder Distribution Volume Histogram (DVH) to toxicities | at 180 days post treatment
  To prospectively correlate dose-volume histograms of the rectum and bladder by studying wall and whole organ volumes to the development of GI and GU toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Niazi, MD, Principal Investigator — Jewish General Hospital
Locations (12):
- Canada (12):
  - Horizon Health Network - Saint John Regional Hospital, Saint John, New Brunswick
  - Complexe hospitalier de la Sagamie, Chicoutimi, Quebec
  - Hôpital de Gatineau, Gatineau, Quebec
  - Hôpital Charles-Lemoyne, Greenfield Park, Quebec
  - Hôpital de la Cité-de-la-santé de Laval, Laval, Quebec
  - CHUM-Notre- Dame, Montreal, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHUQ, L'Hôtel-Dieu de Québec, Québec, Quebec
  - Centre de santé Rimouski-Neigette, Rimouski, Quebec
  - CHUS - Hôpital Fleurimont, Sherbrooke, Quebec
  - Centre Hospitalier régional de Trois-Rivières, Trois-Rivières, Quebec

REFERENCES:
- [Derived] Khriguian J, Tsui JMG, Vaughan R, Kucharczyk MJ, Nabid A, Bettahar R, Vincent L, Martin AG, Jolicoeur M, Yassa M, Barkati M, Igidbashian L, Bahoric B, Archambault R, Villeneuve H, Mohiuddin M, Niazi T. The Clinical Significance of Bone Mineral Density Changes Following Long-Term Androgen Deprivation Therapy in Localized Prostate Cancer Patients. J Urol. 2021 Jun;205(6):1648-1654. doi: 10.1097/JU.0000000000001646. Epub 2021 Feb 12. PMID 33577365